CLINICAL TRIAL: NCT00647621
Title: Steady-State Bioequivalence Study of Extended Phenytoin Sodium Capsules (100 mg; Mylan) and Dilantin® Kapseals® (100 mg; Pfizer) in Healthy Adult Volunteers
Brief Title: Steady-State Study of Extended Phenytoin Sodium Capsules 100 mg and Dilantin® Kapseals® 100 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Will Sullvan, Global Head of Product Risk and Safety Management, Mylan Inc.
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PHEN-0529
Record Dates: First submitted 2008-03-30; First posted 2008-04-01 (Estimated); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Healthy

ARMS (2):
- 1 (Experimental): Extended Phenytoin Sodium Capsules 100 mg
  Interventions: Drug: Extended Phenytoin Sodium Capsules 100 mg
- 2 (Active Comparator): Dilantin® Kapseals® 100 mg
  Interventions: Drug: Dilantin® Kapseals® 100 mg

INTERVENTIONS:
Drug: Extended Phenytoin Sodium Capsules 100 mg — 3x100mg for 14 days, fasting conditions, continuing 2 days with dosing following high-fat breakfast on Day 16
  Arms: 1
Drug: Dilantin® Kapseals® 100 mg — 3x100mg for 14 days, fasting conditions, continuing 2 days with dosing following high-fat breakfast on Day 16
  Arms: 2

SUMMARY:
The objective of this study was to investigate the steady-state bioequivalence of Mylan's extended phenytoin sodium capsules, 100mg (3x100mg), to Pfizer's Dilantin® Kapseals®, 100mg (3x100mg), under both fasting and fed conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years and older.
2. Sex: Male and/or females of non-childbearing potential.

   1. Women will not be considered of childbearing potential if one of the following is reported and documented on the medical history:

      1. postmenopausal with an absence of menses for at least one (1) year, or
      2. bilateral oophorectomy with or without a hysterectomy and an absence of bleeding for at least 6 months, or
      3. total hysterectomy
   2. During the course of the study, from study screen until study exit - including the washout period, men must use a spermicide containing barrier method of contraception. This advice should be documented in the informed consent form.
3. Weight: At least 60 kg (132 lbs) for men and 48 kg (106 lbs) for women and all subjects within 15% of their Ideal Body Weight (IBW), as referenced by the Table of "Desirable Weights of Adults" Metropolitan Life Insurance Company, 1999 (See Part II ADMINISTRATIVE ASPECTS OF BIOEQUIVALENCE PROTOCOLS).
4. All subjects should be judged normal and healthy during a pre-study medical evaluation (physical examination, laboratory evaluation, Hepatitis B and Hepatitis C tests, HIV test, 12-lead ECG, and urine drug screen including amphetamine, barbiturates, benzodiazepines, cannabinoid, cocaine, opiate screen, phencyclidine, and methadone) performed within 21 days of the initial dose of study medication.

Exclusion Criteria:

1. Institutionalized subjects will not be used.
2. Social Habits:

   1. Use of any tobacco-containing products within 1 year of the start of the study.
   2. Ingestion of any alcoholic, caffeine- or xanthine-containing food or beverage within the 48 hours prior to the initial dose of study medication.
   3. Ingestion of any vitamins or herbal products within 7 days prior to the initial dose of the study medication.
   4. Any recent, significant change in dietary or exercise habits.
   5. A positive test for any drug included in the urine drug screen.
   6. History of drug and/or alcohol abuse.
3. Medications:

   1. Use of any prescription or over-the-counter (OTC) medications within the 14 days prior to the initial dose of study medication.
   2. Use of any hormone replacement therapy within 3 months prior to study medication dosing.
   3. Use of any medication known to alter hepatic enzyme activity within 28 days prior to the initial dose of study medication.
4. Diseases:

   1. History of any significant cardiovascular, hepatic, renal, pulmonary, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, or neurologic disease.
   2. Acute illness at the time of either the pre-study medical evaluation or dosing.
   3. A positive HIV, Hepatitis B, or Hepatitis C test.
   4. History of porphyria.
   5. History of diabetes.
5. Abnormal and clinically significant laboratory test results:

   1. Clinically significant deviation from the Guide to Clinically Relevant Abnormalities (See Part II ADMINISTRATIVE ASPECTS OF BIOEQUIVALENCE PROTOCOLS).
   2. Abnormal and clinically relevant ECG tracing.
6. Donation or loss of a significant volume of blood or plasma (> 450 mL) within 28 days prior to the initial dose of study medication.
7. Subjects who have received an investigational drug within 30 days prior to the initial dose of study medication.
8. Allergy or hypersensitivity to phenytoin or any other hydantoins.
9. History of difficulties in swallowing, or any gastrointestinal disease which could affect the drug absorption.
10. Consumption of grapefruit or grapefruit containing products within 7 days of drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2005-10; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: James D Carlson, Pharm. D., Principal Investigator — PRACS Institute Ltd.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States

REFERENCES:
- See also: Mylan Pharmaceuticals Inc. - Clinical Trial Results — http://www.mpibiostudies.com
- See also: Daily Med - posting of most recent submitted labelling to the Food and Drug Administration (FDA) and currently in use — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html